CLINICAL TRIAL: NCT07236814
Title: Suraxavir Marboxil And Oseltamivir for Influenza Prophylaxis Under a Hospital-based Setting
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Bin Cao, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Sur-Ose-Hospital-Prophylaxis
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Influenza
Keywords: influenza; suraxavir marboxil; oseltamivir
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oseltamivir Arm (Experimental): All subjects will be randomized to receive suraxavir marboxil placebo (40mg on the first day) and oseltamivir (75mg each day during the first five days).
  Interventions: Drug: Oseltamivir; Drug: Suraxavir marboxil placebo
- suraxavir marboxil (Experimental): All subjects will be randomized to receive oseltamivir placebo(75mg each day during the first five days) and suraxavir marboxil (40mg on the first day).
  Interventions: Drug: Suraxavir marboxil; Drug: Oseltamivir
- Control Arm (Placebo Comparator): All subjects will be randomized to receive oseltamivir placebo(75mg each day during the first five days) and suraxavir marboxil placebo (40mg on the first day).
  Interventions: Drug: Oseltamivir Placebo; Drug: Suraxavir marboxil placebo

INTERVENTIONS:
Drug: Suraxavir marboxil — Suraxavir marboxil (40mg on the first day)
  Arms: suraxavir marboxil
Drug: Oseltamivir Placebo — Oseltamivir placebo(75mg each day during the first five days)
  Arms: Control Arm
Drug: Oseltamivir — Oseltamivir (75mg each day during the first five days)
  Arms: Oseltamivir Arm; suraxavir marboxil
Drug: Suraxavir marboxil placebo — Suraxavir marboxil placebo (40mg on the first day).
  Arms: Control Arm; Oseltamivir Arm

SUMMARY:
This study aims to evaluate the efficacy of antiviral prophylaxis in preventing in-hospital influenza transmission. We will enroll hospitalized patients with confirmed influenza (index cases) and their uninfected roommates (room contacts). These room contacts will be randomized in a 1:1:1 ratio to one of three prophylactic groups: placebo, suraxavir marboxil, or oseltamivir. The primary outcome will be the rate of influenza infection among the room contacts, which will be monitored to determine the effectiveness of the interventions.

ELIGIBILITY:
1.Inclusion Criteria:

(1)Inclusion Criteria for Index Cases:

① Patients hospitalized at a participating medical institution.

* The subject and/or their legal guardian agrees to participate in this clinical study, has signed the informed consent form, and is able to comply with the protocol requirements for follow-up and complete all study procedures and assessments.

  * Age ≥ 2 years.

    * Positive for influenza virus as determined by a Rapid Antigen Test (RAT) or Nucleic Acid Amplification Test (NAAT) on a respiratory specimen (e.g., oropharyngeal swab, nasopharyngeal swab, sputum, or bronchoalveolar lavage fluid).

      (2) Inclusion Criteria for Room Contacts:

      ① Patients hospitalized at a participating medical institution.
* The subject and/or their legal guardian agrees to participate in this clinical study, has signed the informed consent form, and is able to comply with the protocol requirements for follow-up and complete all study procedures and assessments.

  ③ Age ≥ 12 years.
  * Expected to remain hospitalized for ≥ 72 hours.

    * Shares a room with at least one hospitalized index case who has been confirmed with influenza virus infection by RAT or NAAT on a respiratory specimen within the last 120 hours and developed influenza-related symptoms within the last 120 hours, and is expected to share the same room for ≥ 24 hours.

      ⑥ Negative for influenza virus as determined by a Nucleic Acid Amplification Test (NAAT) on a throat swab collected on Day 1.

      3.Exclusion Criteria

      (1) Index Cases There are no exclusion criteria for index cases. (2) Exclusion Criteria for Room Contacts:
      * Room contacts with a known allergy to the active ingredients or excipients of the investigational drugs.
* Room contacts who have been diagnosed with or have had an influenza virus infection in the past 12 weeks.

  * Use of any anti-influenza antiviral drugs within 2 weeks prior to screening, including: neuraminidase inhibitors, polymerase inhibitors, hemagglutinin inhibitors, and M2 ion channel blockers (e.g., Oseltamivir, Zanamivir, Peramivir, Favipiravir, Arbidol, Baloxavir Marboxil, Amantadine, or Rimantadine, or other anti-influenza drugs approved by the NMPA).

    * Known to be pregnant or breastfeeding. (Subjects who suspect they may be pregnant must report this to the investigator, who will confirm with a pregnancy test).

      * History of fever (axillary temperature ≥ 37.3°C) within 72 hours prior to screening.

        * Child-Pugh class B or C, or an eGFR ≤ 60 mL·min-¹·(1.73 m²)-¹. ⑦ Any subject deemed unsuitable for participation in the study by the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-06 (Estimated)

PRIMARY OUTCOMES:
The proportion of room contacts who develop clinical influenza within 5 days, with a virus subtype consistent with that of the index case. | within 5 days
  The proportion of room contacts who develop clinical influenza* within 5 days, with a virus subtype consistent with that of the index case.
  *Clinical influenza is defined as a positive influenza virus detection by Rapid Antigen Test (RAT) or Nucleic Acid Amplification Test (NAAT), accompanied by at least one respiratory symptom (fever or chills, muscle or joint pain, headache, fatigue) and at least onesystemic symptom (cough, nasal congestion, sore throat).

SECONDARY OUTCOMES:
The proportion of room contacts who develop clinical influenza (as defined above) within 10 days | within 10 days
  The proportion of room contacts who develop clinical influenza (as defined above) within 10 days, with a virus subtype consistent with that of the index case.
The proportion of room contacts with laboratory-confirmed influenza within 5 days | Within 5 days
  The proportion of room contacts with laboratory-confirmed influenza (defined as a positive influenza virus RAT or NAAT result, regardless of symptoms) within 5 days, with a virus subtype consistent with that of the index case.
The incidence of post-treatment changes in the influenza virus sequence | Within 10 days
  Among room contacts who become infected with influenza virus within 10 days, the incidence of post-treatment changes in the influenza virus sequence (based on viral sequence analysis). This includes the incidence of events such as the I38T amino acid substitution, the H275Y amino acid substitution, and other emerging amino acid substitutions in the PA and NA sequences.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship hospital, Beijing, Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No